CLINICAL TRIAL: NCT04232670
Title: Pancreatic Endotherapy for Refractory Chronic Pancreatitis
Acronym: PERCePT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gregory Cote, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00087299
Record Dates: First submitted 2019-12-06; First posted 2020-01-18 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Duct Stone; Pancreatic Duct Stricture; Pancreatic Duct Dilatation
Keywords: pancreas; pancreatic duct; ductal stone; duct stricture; ERCP; pancreatic duct obstruction; duct calcification
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: In addition to the participant and the investigator assessing outcomes, study coordinators involved in collecting outcomes data will be masked to the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS + SHAM (Sham Comparator): All subjects will undergo anesthesia administered sedation and endoscopic ultrasound (EUS). The endoscopist will assess the pancreas for parenchymal and ductal features of chronic pancreatitis and confirm the absence of exclusion criteria (such as the presence of an occult pancreatobiliary malignancy).
  Interventions: Procedure: EUS + SHAM
- EUS + Pancreatic Endotherapy (Experimental): If randomized to ERCP with pancreatic endotherapy, the endoscopist will proceed with this intervention immediately following the completion of EUS and treatment allocation (during the same anesthesia). Pancreatic endotherapy may include any or all of the following maneuvers: pancreatic endoscopic sphincterotomy, stricture dilation using a bougie or hydrostatic balloon catheter, pancreatic stone extraction with or without mechanical or electrohydraulic lithotripsy, extracorporeal shock wave lithotripsy, and stent placement. Overall technical success will be defined by the ability to insert at least one pancreatic stent across the dominant main pancreatic duct obstruction. Technical success for pancreatic stone treatment will be defined by the ability to remove all fluoroscopically visible main pancreatic duct stones.
  Interventions: Procedure: EUS + Pancreatic Endotherapy

INTERVENTIONS:
Procedure: EUS + SHAM — Endoscopic Ultrasound
  Arms: EUS + SHAM
Procedure: EUS + Pancreatic Endotherapy — Pancreatic endotherapy may include any or all of the following maneuvers: pancreatic endoscopic sphincterotomy, stricture dilation using a bougie or hydrostatic balloon catheter, pancreatic stone extraction with or without mechanical or electrohydraulic lithotripsy, extracorporeal shock wave lithotripsy, and stent placement.
  Arms: EUS + Pancreatic Endotherapy

SUMMARY:
The purpose of this study is to evaluate whether endoscopic ultrasound (EUS) only versus EUS + endoscopic retrograde cholangiopancreatography (ERCP) with pancreatic endotherapy reduces pain in the treatment of chronic pancreatitis with pancreatic duct obstruction.

DETAILED DESCRIPTION:
This is a single center, pilot, sham-controlled clinical trial of ERCP with pancreatic endotherapy for pain secondary to chronic calcific pancreatitis with main pancreatic duct obstruction. Potential subjects will undergo a comprehensive baseline assessment including Quantitative Sensory Testing, to ensure enrollment criteria are met and baseline covariates are measured. Eligible subjects will complete a 14-day run-in period. If eligibility criteria persist, subjects will be randomized to diagnostic endoscopic ultrasound (EUS) + sham pancreatic endotherapy or diagnostic EUS + ERCP with pancreatic endotherapy as defined in the study protocol. Subjects will be followed by a blinded physician for the next 90 days, at which time the pilot trial outcomes will be measured. Regardless of outcomes, all subjects will be followed longitudinally for 12 months after randomization.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years
* Main pancreatic duct obstruction, defined by the presence of one or both of the following features:
* Main pancreatic duct calcification with upstream main duct dilation ≥6mm.
* Main pancreatic duct stricture, defined by the presence of main pancreatic duct narrowing with upstream main duct dilation ≥6mm.
* Baseline average abdominal pain score ≥4 during the run-in period, based on Ecological Momentary Assessment 11-point Numeric Rating Scale
* Ability to provide written, informed consent

Exclusion Criteria

* Symptoms attributable to a pancreatic pseudocyst or walled off necrosis
* Clinical suspicion of pancreatobiliary malignancy*
* Low probability of follow-up to complete study objectives
* Pregnancy or incarceration
* Medical comorbidities that contraindicate the performance of ERCP
* Previous pancreatic endotherapy
* Current Opioid Misuse Measure score ≥9
* Does not have access to a mobile phone * Pancreatobiliary malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Cote, MD, MS, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- EUS + Pancreatic Endotherapy: If randomized to endoscopic retrograde cholangiopancreatography (ERCP) with pancreatic endotherapy, the endoscopist will proceed with this intervention immediately following the completion of EUS and treatment allocation (during the same anesthesia). Pancreatic endotherapy may include any or all of the following maneuvers: pancreatic endoscopic sphincterotomy, stricture dilation using a bougie or hydrostatic balloon catheter, pancreatic stone extraction with or without mechanical or electrohydraulic lithotripsy, extracorporeal shock wave lithotripsy, and stent placement. Overall technical success will be defined by the ability to insert at least one pancreatic stent across the dominant main pancreatic duct obstruction. Technical success for pancreatic stone treatment will be defined by the ability to remove all fluoroscopically visible main pancreatic duct stones.
  EUS + Pancreatic Endotherapy: Pancreatic endotherapy may include any or all of the following maneuvers: pancreatic endoscopic sphincterotomy, stricture dilation using a bougie or hydrostatic balloon catheter, pancreatic stone extraction with or without mechanical or electrohydraulic lithotripsy, extracorporeal shock wave lithotripsy, and stent placement.
Period: Overall Study
Arm/Group | EUS + SHAM | EUS + Pancreatic Endotherapy
Started | 6 | 8
Completed | 5 | 8
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EUS + SHAM | EUS + Pancreatic Endotherapy | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 0 | 1 | 1
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [37 to 79] | 46.5 [27 to 66] | 53 [33 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Average Daily Pain Score on the Numeric Rating Scale
Description: The percent change in average daily pain score from the daily diaries during the 14-day period preceding the 90-day assessment, compared to the average daily pain reported during the 14-day run-in. The investigators employed the standardized 11-point Numeric Rating Scale (NRS) to capture average daily pain with the empirically-supported anchors of 0=No Pain and 10=Worst Pain Imaginable.
Time Frame: Day -14 to Day 90
Population: The analysis population is the 9 participants who completed the Ecological Momentary Assessment (EMA) at both the start of the study and at the 90-day follow-up.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | EUS + SHAM | EUS + Pancreatic Endotherapy
Number analyzed (Participants) | 4 | 5
Percent Change | -36.6 [-39.3 to -11.6] | -53.7 [-100.0 to -27.9]

ADVERSE EVENTS:
Time Frame: An Adverse Event form was used to document reportable adverse events (AEs) for this study, which included: 1. All non-serious adverse events related to abdominal pain in addition to all serious adverse events were reported through Day 30 2. All serious adverse events (SAEs) were reported through the end of study (12 months post randomization) 3. All acute pancreatitis events or pancreatitis-related pain events that occur were reported through end of study ((12 months post randomization).
Description: Unblinded personnel reported AEs between randomization and Day 30. Blinded personnel reported AEs between Day 30 post randomization & up to the 90 day visit, then unblinded personnel reported any SAEs at Day 90 and afterwards.
Arm/Group | EUS + SHAM | EUS + Pancreatic Endotherapy
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 4/6 | 6/8
Other Adverse Events (participants affected / at risk) | 0/6 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EUS + SHAM (N=6) | EUS + Pancreatic Endotherapy (N=8)
Acute pancreatitis > 30 days from randomization (Hepatobiliary disorders) | 2 (8) | 2 (2)
Acute pancreatitis within 30 days of randomization (Hepatobiliary disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (6) | 4 (14)
Chronic pancreatitis (Hepatobiliary disorders) | 3 (4) | 2 (3)
Acute pain (General disorders) | 0 (0) | 1 (1)
Post procedural pain (Gastrointestinal disorders) | 1 (1) | 1 (2)
Active Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Anaphylaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Elevated liver enzyme levels (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Suprapubic pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Temporal headache (General disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EUS + SHAM (N=6) | EUS + Pancreatic Endotherapy (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Small sample size due to recruitment challenges

- It is difficult to recruit for the sham arm because endotherapy is widely utilized in clinical practice and advocated by expert consensus. Patients with painful chronic pancreatitis are disabled by their disease and often keen to try something even when risks are fixed and benefit unpredictable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT04232670/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT04232670/ICF_000.pdf